CLINICAL TRIAL: NCT01935791
Title: Investigating Brown Adipose Tissue Activation in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 13HH0688
Record Dates: First submitted 2013-07-25; First posted 2013-09-05 (Estimated); Results first posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Metabolic Diseases
Keywords: Metabolic Diseases
MeSH Terms: conditions — Metabolic Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Period 1 Visit 1 - Cold PET-CT Vehicle, Visit 2 -Warm PET-CT Vehicle (Active Comparator): Visit 1. Participants underwent F-fluorodeoxyglucose (18F-FDG) positron emission tomography, computerised tomography-(PET)CT, whilst wearing a cooling vest and receiving an infusion of gelofusine.
  Visit 2 Participants underwent F-fluorodeoxyglucose (18F-FDG) positron emission tomography, computerised tomography-(PET)CT, whilst receiving an infusion of gelofusine without a cooling vest.
  Interventions: Other: Period 1 Visit 1 - Cold PET-CT Vehicle, Visit 2 -Warm PET-CT Vehicle
- Period 1 Visit 1 - Cold PET-CT Vehicle, Visit 2 -Warm PET-CT Glucagon (Experimental): Visit 1. Participants underwent F-fluorodeoxyglucose (18F-FDG) positron emission tomography, computerised tomography-(PET)CT, whilst wearing a cooling vest and receiving an infusion of gelofusine Visit 2 Participants underwent F-fluorodeoxyglucose (18F-FDG) positron emission tomography, computerised tomography-(PET)CT, whilst receiving an infusion of Glucagon at a dose of 50ng/kg/min without a cooling vest.
  Interventions: Drug: Period 1 Visit 1 - Cold PET-CT Vehicle, Visit 2 -Warm PET-CT Glucagon
- Period 1 Visit 1 - Cold PET-CT Vehicle, no visit 2 as BAT negative (Active Comparator): Visit 1. Participants underwent F-fluorodeoxyglucose (18F-FDG) positron emission tomography, computerised tomography-(PET)CT, whilst wearing a cooling vest and receiving an infusion of gelofusine.
  No brown adipose tissue (BAT) identified on visit 1, therefore no visit 2.
  Interventions: Other: Period 1 Visit 1 - Cold PET-CT Vehicle, no visit 2 as BAT negative
- Period 2 - Visit 1 Warm Control vehicle, Visit 2 Warm Glucagon, Visit 3 Cold control (Experimental): Visit 1- Each participant had calorimetry testing and thermal imaging whilst receiving an infusion of gelofusine. They were situated in an ambient temperature of 22-25 degrees celsius.
  Visit 2 - Each participant had calorimetry testing and thermal imaging whilst receiving an infusion of Glucagon at a dose of 50ng/kg/min. They were situated in an ambient temperature of 22-25 degrees celsius. Visit 3 - Each participant had calorimetry testing and thermal imaging whilst receiving an infusion of gelofusine and wearing a cooling vest.
  Interventions: Drug: Period 2 - Visit 1 Warm Control vehicle, Visit 2 Warm Glucagon, Visit 3 Cold control
- Period 2 - Visit 1 Warm Glucagon, Visit 2 Cold control , Visit 3 Warm control (Experimental): Visit 1- Each participant had calorimetry testing and thermal imaging whilst receiving an infusion of Glucagon at a dose of 50ng/kg/min. They were situated in an ambient temperature of 22-25 degrees celsius.
  Visit 2 - Each participant had calorimetry testing and thermal imaging whilst receiving an infusion of gelofusine and wearing a cooling vest.
  Visit 3 Each participant had calorimetry testing and thermal imaging whilst receiving an infusion of gelofusine. They were situated in an ambient temperature of 22-25 degrees celsius.
  Interventions: Drug: Period 2 - Visit 1 Warm Glucagon, Visit 2 Cold control , Visit 3 Warm control
- Period 2 -Visit 1 cold control, Visit 2 warm control, Visit 3 Warm glucagon (Experimental): Visit 1 - Each participant had calorimetry testing and thermal imaging whilst receiving an infusion of gelofusine and wearing a cooling vest.
  Visit 2 - Each participant had calorimetry testing and thermal imaging whilst receiving an infusion of gelofusine. They were situated in an ambient temperature of 22-25 degrees celsius.
  Visit 3 - Each participant had calorimetry testing and thermal imaging whilst receiving an infusion of Glucagon at a dose of 50ng/kg/min. They were situated in an ambient temperature of 22-25 degrees celsius.
  Interventions: Drug: Period 2 -Visit 1 cold control, Visit 2 warm control, Visit 3 Warm glucagon
- Period 2 -Visit 1 cold control, visit 2 warm glucagon, visit 3 warm control (Experimental): Visit 1 - Each participant had calorimetry testing and thermal imaging whilst receiving an infusion of gelofusine and wearing a cooling vest.
  Visit 2- Each participant had calorimetry testing and thermal imaging whilst receiving an infusion of Glucagon at a dose of 50ng/kg/min. They were situated in an ambient temperature of 22-25 degrees Celsius.
  Visit 3 - Each participant had calorimetry testing and thermal imaging whilst receiving an infusion of gelofusine. They were situated in an ambient temperature of 22-25 degrees Celsius.
  Interventions: Drug: Period 2 -Visit 1 cold control, visit 2 warm glucagon, visit 3 warm control
- Period 2- Visit 1 Warm glucagon, visit 2 warm control, visit 3 cold control (Experimental): Visit 1- Each participant had calorimetry testing and thermal imaging whilst receiving an infusion of Glucagon at a dose of 50ng/kg/min. They were situated in an ambient temperature of 22-25 degrees Celsius.
  Visit 2 Each participant had calorimetry testing and thermal imaging whilst receiving an infusion of gelofusine. They were situated in an ambient temperature of 22-25 degrees Celsius.
  Visit 3- Each participant had calorimetry testing and thermal imaging whilst receiving an infusion of gelofusine and wearing a cooling vest.
  Interventions: Drug: Period 2- Visit 1 Warm glucagon, visit 2 warm control, visit 3 cold control
- Period 2 - Visit 1 Warm control, visit 2 cold control, visit 3 warm glucagon (Experimental): Visit 1 Each participant had calorimetry testing and thermal imaging whilst receiving an infusion of gelofusine. They were situated in an ambient temperature of 22-25 degrees Celsius.
  Visit 2- Each participant had calorimetry testing and thermal imaging whilst receiving an infusion of gelofusine and wearing a cooling vest.
  Visit 3 Each participant had calorimetry testing and thermal imaging whilst receiving an infusion of Glucagon at a dose of 50ng/kg/min. They were situated in an ambient temperature of 22-25 degrees Celsius
  Interventions: Drug: Period 2 - Visit 1 Warm control, visit 2 cold control, visit 3 warm glucagon

INTERVENTIONS:
Other: Period 1 Visit 1 - Cold PET-CT Vehicle, Visit 2 -Warm PET-CT Vehicle — Temperature
  Arms: Period 1 Visit 1 - Cold PET-CT Vehicle, Visit 2 -Warm PET-CT Vehicle
Drug: Period 1 Visit 1 - Cold PET-CT Vehicle, Visit 2 -Warm PET-CT Glucagon — Hormone
  Arms: Period 1 Visit 1 - Cold PET-CT Vehicle, Visit 2 -Warm PET-CT Glucagon
Other: Period 1 Visit 1 - Cold PET-CT Vehicle, no visit 2 as BAT negative — Temperature
  Arms: Period 1 Visit 1 - Cold PET-CT Vehicle, no visit 2 as BAT negative
Drug: Period 2 - Visit 1 Warm Control vehicle, Visit 2 Warm Glucagon, Visit 3 Cold control — Hormone
  Arms: Period 2 - Visit 1 Warm Control vehicle, Visit 2 Warm Glucagon, Visit 3 Cold control
Drug: Period 2 - Visit 1 Warm Glucagon, Visit 2 Cold control , Visit 3 Warm control — Hormone
  Arms: Period 2 - Visit 1 Warm Glucagon, Visit 2 Cold control , Visit 3 Warm control
Drug: Period 2 -Visit 1 cold control, Visit 2 warm control, Visit 3 Warm glucagon — hormone
  Arms: Period 2 -Visit 1 cold control, Visit 2 warm control, Visit 3 Warm glucagon
Drug: Period 2 -Visit 1 cold control, visit 2 warm glucagon, visit 3 warm control — hormone
  Arms: Period 2 -Visit 1 cold control, visit 2 warm glucagon, visit 3 warm control
Drug: Period 2- Visit 1 Warm glucagon, visit 2 warm control, visit 3 cold control — hormone
  Arms: Period 2- Visit 1 Warm glucagon, visit 2 warm control, visit 3 cold control
Drug: Period 2 - Visit 1 Warm control, visit 2 cold control, visit 3 warm glucagon — Hormone
  Arms: Period 2 - Visit 1 Warm control, visit 2 cold control, visit 3 warm glucagon

SUMMARY:
The purpose of this study is to determine what can activate brown adipose tissue (BAT).

DETAILED DESCRIPTION:
We will investigate different stimuli (i.e. hormones) to determine which can stimulate BAT.

ELIGIBILITY:
Inclusion Criteria:

* aged >18 years

Exclusion Criteria:

* medical conditions
* recreational drug use
* participation in other trials within the preceding 2 months
* blood donation within 3 months of study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-07; Primary Completion 2018-11-05 (Actual); Study Completion 2018-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Waljit Dhillo, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Salem V, Izzi-Engbeaya C, Coello C, Thomas DB, Chambers ES, Comninos AN, Buckley A, Win Z, Al-Nahhas A, Rabiner EA, Gunn RN, Budge H, Symonds ME, Bloom SR, Tan TM, Dhillo WS. Glucagon increases energy expenditure independently of brown adipose tissue activation in humans. Diabetes Obes Metab. 2016 Jan;18(1):72-81. doi: 10.1111/dom.12585. Epub 2015 Nov 20. PMID 26434748
- See also: Thermal Imaging Is a Noninvasive Alternative to PET/CT for Measurement of Brown Adipose Tissue Activity in Humans — http://jnm.snmjournals.org/content/59/3/516.long

RESULTS

PARTICIPANT FLOW:
Groups:
- Period 2 -Visit 1 Warm Control, Visit 2 Cold Control, Visit 3 Warm Glucagon: Visit 1 Each participant had calorimetry testing and thermal imaging whilst receiving an infusion of gelofusine. They were situated in an ambient temperature of 22-25 degrees Celsius.
  Visit 2- Each participant had calorimetry testing and thermal imaging whilst receiving an infusion of gelofusine and wearing a cooling vest.
  Visit 3 Each participant had calorimetry testing and thermal imaging whilst receiving an infusion of Glucagon at a dose of 50ng/kg/min. They were situated in an ambient temperature of 22-25 degrees Celsius
Period: Period 1
Arm/Group | Period 1 Visit 1 - Cold PET-CT Vehicle, Visit 2 -Warm PET-CT Vehicle | Period 1 Visit 1 - Cold PET-CT Vehicle, Visit 2 -Warm PET-CT Glucagon | Period 1 Visit 1 - Cold PET-CT Vehicle, no Visit 2 as BAT Negative | Period 2 - Visit 1 Warm Control Vehicle, Visit 2 Warm Glucagon, Visit 3 Cold Control | Period 2 - Visit 1 Warm Glucagon, Visit 2 Cold Control , Visit 3 Warm Control | Period 2 -Visit 1 Cold Control, Visit 2 Warm Control, Visit 3 Warm Glucagon | Period 2 -Visit 1 Cold Control, Visit 2 Warm Glucagon, Visit 3 Warm Control | Period 2- Visit 1 Warm Glucagon, Visit 2 Warm Control, Visit 3 Cold Control | Period 2 -Visit 1 Warm Control, Visit 2 Cold Control, Visit 3 Warm Glucagon
Started | 4 | 4 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 4 | 4 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Period 1 Visit 1 - Cold PET-CT Vehicle, Visit 2 -Warm PET-CT Vehicle | Period 1 Visit 1 - Cold PET-CT Vehicle, Visit 2 -Warm PET-CT Glucagon | Period 1 Visit 1 - Cold PET-CT Vehicle, no Visit 2 as BAT Negative | Period 2 - Visit 1 Warm Control Vehicle, Visit 2 Warm Glucagon, Visit 3 Cold Control | Period 2 - Visit 1 Warm Glucagon, Visit 2 Cold Control , Visit 3 Warm Control | Period 2 -Visit 1 Cold Control, Visit 2 Warm Control, Visit 3 Warm Glucagon | Period 2 -Visit 1 Cold Control, Visit 2 Warm Glucagon, Visit 3 Warm Control | Period 2- Visit 1 Warm Glucagon, Visit 2 Warm Control, Visit 3 Cold Control | Period 2 -Visit 1 Warm Control, Visit 2 Cold Control, Visit 3 Warm Glucagon
Started | 0 | 0 | 0 | 2 | 3 | 1 | 1 | 3 | 1
Completed | 0 | 0 | 0 | 2 | 3 | 1 | 1 | 3 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants who were randomised
Arm/Group | All Participants
Number analyzed (Participants) | 11
Age, Continuous [Mean (Full Range); unit: years] | 26 [20 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants] — All participants were recruited from the Greater London area in England
  Participants
    United Kingdom | 11
BMI [Mean (Full Range); unit: kg/m2] | 22.5 [20.5 to 25.2]

OUTCOME MEASURES:

1. Primary Outcome: Brown Adipose Tissue Activation Following Glucagon or Saline Infusion
Description: Period 1 Brown Adipose Tissue (BAT) activation measured using metabolic rate of glucose (MR[gluc]) during F-fluorodeoxyglucose (18F-FDG) positron emission tomography (PET-CT) for Cold PET-CT Vehicle vs Warm PET-CT Vehicle vs warm PET-CT Glucagon.
Time Frame: 2hours
Population: Period 1 Parallel design (3 out of 11 participants did not have BAT activation and therefore they were not included in the analysis).
  Period 2 Crossover design
Measure: Mean (Standard Deviation); unit: MR[gluc] umol/kg/min
Groups:
- Period 1 Cold PET-CT Vehicle: Visit 1. emission tomography, computerised tomography-(PET)CT, whilst wearing a cooling vest and receiving an infusion of gelofusine.
- Period 1 Warm PET-CT Vehicle: Participants underwent F-fluorodeoxyglucose (18F-FDG) positron emission tomography, computerised tomography-(PET)CT, whilst receiving an infusion of gelofusine without a cooling vest.
- Period 1 Warm PET(CT) Glucagon: Participants underwent F-fluorodeoxyglucose (18F-FDG) positron emission tomography, computerised tomography-(PET)CT, whilst receiving an infusion of Glucagon at a dose of 50ng/kg/min without a cooling vest.
Arm/Group | Period 1 Cold PET-CT Vehicle | Period 1 Warm PET-CT Vehicle | Period 1 Warm PET(CT) Glucagon
Number analyzed (Participants) | 8 | 4 | 4
MR[gluc] umol/kg/min | 0.074 (0.007) | 0.010 (0.003) | 0.029 (0.008)
Statistical Analysis 1: Comparison: Period 1 Cold PET-CT Vehicle vs Period 1 Warm PET-CT Vehicle vs Period 1 Warm PET(CT) Glucagon; Test type: Other; p < 0.01, ANOVA — The p-values were adjusted for multiple comparisons. The a priori threshold for statistical significance is p<0.05; plus Tukey test

2. Primary Outcome: Increase in Energy Expenditure Following Glucagon or Saline Infusion
Description: Period 2 Increase in energy expenditure measured using indirect calorimetry for Cold control vs Warm Control vs Warm Glucagon.
Time Frame: 2hours
Population: Period 2 Crossover design
Measure: Mean (Standard Deviation); unit: increase in energy expenditure kcal/day
Groups:
- Period 2 - Cold Control: Each participant had calorimetry testing and thermal imaging whilst receiving an infusion of gelofusine and wearing a cooling vest.
- Period 2 - Warm Control: Each participant had calorimetry testing and thermal imaging whilst receiving an infusion of gelofusine. They were situated in an ambient temperature of 22-25 degrees celsius.
- Period 2 -Warm Glucagon: Each participant had calorimetry testing and thermal imaging whilst receiving an infusion of Glucagon at a dose of 50ng/kg/min. They were situated in an ambient temperature of 22-25 degrees celsius.
Arm/Group | Period 2 - Cold Control | Period 2 - Warm Control | Period 2 -Warm Glucagon
Number analyzed (Participants) | 11 | 11 | 11
increase in energy expenditure kcal/day | 193.0 (27.2) | 41.1 (70) | 230.8 (30.1)
Statistical Analysis 1: Comparison: Period 2 - Cold Control vs Period 2 - Warm Control vs Period 2 -Warm Glucagon; Test type: Other; p < 0.001, ANOVA; plus Tukey test

ADVERSE EVENTS:
Time Frame: 3 years
Description: Patients were monitored for adverse events throughout each visit and had the contact details of the main investigator for any issues in between visits.
Groups:
- Period 1 Visit 1 Cold Vehicle: Participants underwent F-fluorodeoxyglucose (18F-FDG) positron emission tomography, computerised tomography-(PET)CT, whilst wearing a cooling vest and receiving an infusion of gelofusine.
- Period 1 Visit 2 Warm Glucagon: Participants underwent F-fluorodeoxyglucose (18F-FDG) positron emission tomography, computerised tomography-(PET)CT, whilst receiving an infusion of Glucagon at a dose of 50ng/kg/min without a cooling vest.
- Period 1 Visit 2 Warm Vehicle: Participants underwent F-fluorodeoxyglucose (18F-FDG) positron emission tomography, computerised tomography-(PET)CT, whilst receiving an infusion of gelofusine without a cooling vest.
- Period 2 Cold Control: Each participant had calorimetry testing and thermal imaging whilst receiving an infusion of gelofusine and wearing a cooling vest.
- Period 2 Warm Control: Each participant had calorimetry testing and thermal imaging whilst receiving an infusion of gelofusine. They were situated in an ambient temperature of 22-25 degrees celsius.
- Period 2 Warm Glucagon: Each participant had calorimetry testing and thermal imaging whilst receiving an infusion of Glucagon at a dose of 50ng/kg/min. They were situated in an ambient temperature of 22-25 degrees celsius.
Arm/Group | Period 1 Visit 1 Cold Vehicle | Period 1 Visit 2 Warm Glucagon | Period 1 Visit 2 Warm Vehicle | Period 2 Cold Control | Period 2 Warm Control | Period 2 Warm Glucagon
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/4 | 0/4 | 0/11 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/4 | 0/4 | 0/11 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/4 | 0/4 | 0/11 | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2014-05-29): https://cdn.clinicaltrials.gov/large-docs/91/NCT01935791/Prot_000.pdf
  • Statistical Analysis Plan (2014-05-29): https://cdn.clinicaltrials.gov/large-docs/91/NCT01935791/SAP_001.pdf